CLINICAL TRIAL: NCT03248999
Title: Determination of the Prevalence of ESBL-producing Enterobacteriaceae as Carbapenem-resistant Enterobacteriaceae in Nursing Homes in Franche-Comté (France).
Brief Title: Prevalence of ESBL-producing Enterobacteriaceae as Carbapenem-resistant Enterobacteriaceae in Nursing Homes.
Acronym: R'EHPAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P/2017/315
Record Dates: First submitted 2017-08-02; First posted 2017-08-15 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-03

CONDITIONS: Drug Resistance, Bacterial
Keywords: multidrug resistance; nursing home; ESBL; CRE

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): realization of a rectal swab or stool sample for all the résidents included in the study.
  Interventions: Diagnostic Test: rectal swab

INTERVENTIONS:
Diagnostic Test: rectal swab — stool samples by rectal swab

SUMMARY:
This study evaluates individual and collective factors of ESBL and CRE carriage in nursing homes.

DETAILED DESCRIPTION:
Epimiological data concerning ESBL an CRE, may differ between nursing home and hospital or community but poor data are available.

Multi-drug resistant bacteria carriage is associated with individual and collective factors wich have to be defined in nursing homes.

ELIGIBILITY:
Inclusion Criteria:

* voluntary residents present in the institution on the study day

Exclusion Criteria:

* dement-wandering resident
* unlikely to cooperate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
ESBL and CRE carriage | the day of the study
  number of residents colonized with a extented-spectrum beta-lactamase-producing Enterobacteriaceae (ESBL) or carbapenem-resistant Enterobacteriaceae (CRE)

SECONDARY OUTCOMES:
patient and establishment factors associated with ESBL and CRE carriage with a questionnaire | the day of the study
  evaluation of risk factors associated with ESBL and CRE carriage and disseminationwith a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Céline C Bouvier-Slekovec, Dr, Principal Investigator — CHU de Besançon
Locations (1):
- CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No